CLINICAL TRIAL: NCT00569517
Title: The Effect of Brief Group Cognitive Behavioral Therapy on Decreasing Metabolic Syndrome Risk Factors in Obese Patients Treated With Atypical Antipsychotics
Brief Title: Cognitive Behavioral Therapy for Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Aljurdi, Rayan - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-21955; 07K19.H
Record Dates: First submitted 2007-12-05; First posted 2007-12-07 (Estimated); Last update posted 2009-03-20 (Estimated); Status verified 2009-03

CONDITIONS: Obesity
Keywords: obesity; CBT; Atypical antipsychotics; metabolic syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 6-CBT-sessions for weight loss
  Interventions: Behavioral: CBT
- 2 (Experimental): Single educational intervention for weight
  Interventions: Other: educational

INTERVENTIONS:
Behavioral: CBT — 6-CBT based sesions
  Arms: 1
Other: educational — subjects receive one hour of nutrition education and 5 weekly phone calls
  Arms: 2

SUMMARY:
The purpose of this pilot study is to assess patient accessibility, interest and response in order to design an adequately powered study to compare brief, group cognitive behavioral therapy (CBT) for weight loss to usual care in non-demented patients above the age of 18 years old who are currently taking atypical antipsychotic medications. This pilot study is necessary, with current limitations of data in this area, to design an adequately powered study to address the difficulties managing metabolic syndrome risk factors in patients on antipsychotics.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and above
2. Patients with diagnosis of schizophrenia, schizoaffective disorder or bipolar disorder determined by assessment with chart review, currently taking at least one atypical antipsychotic, started at least 2 months prior to randomization
3. Body Mass Index (BMI) greater than 30
4. ability to consent to treatment, determined by the patient's treating/referring physician

Exclusion Criteria:

1. Patients with premorbid medical problems that preclude involvement in a weight loss program
2. Active substance abuse or dependence, indicated by a positive urine drug screen in the last 3 months
3. Mini- Mental Status Exam (MMSE) less than 24
4. active psychosis or mania, determined by administration of the PANSS score greater than 3 on the following items; delusions, conceptual disorganization, hallucinatory behavior, blunted affect, social withdrawal, lack of spontaneity and conversation flow, mannerisms and posturing, and unusual thought content, and YMRS greater than 10, respectively
5. active major depressive episode, determined by administration of HAM-D greater than 13
6. patients taking any medications for weight loss or currently enrolled in a weight loss program
7. changes in medication regimen for diabetes or dyslipidemia within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The accessibility to overweight outpatients with stable psychotic or mood disorders, currently treated with atypical antipsychotics willing to participate in a research study involving CBT. | 3 months

SECONDARY OUTCOMES:
Measure outcome parameters; body mass index, total cholesterol, low-density lipoproteins, triglycerides, fasting blood sugar, waist circumference, blood pressure & pulse among patients receiving CBT treatment or usual care at baseline, 6 wks & 12 wks. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Rayan Aljurdi, MD, Principal Investigator — Michael E. DeBakey VA Medical Center (152)
Locations (1):
- Michael E. DeBakey VA Medical Center (152), Houston, Texas, United States